CLINICAL TRIAL: NCT00783380
Title: Double Blind Randomized Comparison of a Subunit- and a Virosomal Influenza Vaccine in Immunocom-Promized Patients
Brief Title: Influenza Vaccination in Immunocompromized Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Boehringer Ingelheim (Industry); Abbott (Industry); Merck Sharp & Dohme LLC (Industry); Solvay Pharmaceuticals (Industry)
Responsible Party: Evison John, MD Oberarzt, Universitätsklinik für Infektiologie, PKT 2B, Inselspital, 3011 Bern, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KEK No 805 (EK 151/03)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Immunosuppression
Keywords: Influenza vaccination; Subunit; Virosomal; HIV/AIDS; Renal Dialysis; Kidney transplantation; Rheumatologic diseases; Immunogenicity; Reactogenicity
MeSH Terms: conditions — Influenza, Human; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virosomal influenza vaccine (Experimental)
  Interventions: Biological: Virosomal influenza vaccine
- Subunit influenza vaccine (Active Comparator)
  Interventions: Biological: Subunit influenza vaccine

INTERVENTIONS:
Biological: Virosomal influenza vaccine — Influvacplus 2005/2006, Solvay Pharma AG, Bern, Switzerland Assigned to all 4 groups if immunocompromized patients
  Arms: Virosomal influenza vaccine
Biological: Subunit influenza vaccine — Influvac 2005/2006, Solvay Pharma AG, Bern, Switzerland Assigned to all 4 groups if immunocompromized patients
  Arms: Subunit influenza vaccine

SUMMARY:
Evaluation of the immunogenicity and reactogenicity of two different formulations of commercially avail-able influenza vaccines in 4 different groups of immunocompromized outpatients (HIV positive patients, patients suffering from rheumatologic diseases and receiving treatment with immunosuppressive drugs and patients undergoing hemodialysis or continuous ambulatory peritoneal dialysis). The aim of the study was to investigate if the newest formulation of influenza vaccines (virosomal vaccines) offer a benefit in immunocompromized patients in comparison to an older subunit formulation.

DETAILED DESCRIPTION:
The infection with influenza is associated with higher morbidity and mortality in risk groups including immunocompromized patients. The virosomal influenza vaccines have been associated with improved immunogenicity in former trials. No direct comparison with older formulations has been conducted so far.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients treated at the Inselspital Bern for:
* HIV infection
* rheumatologic diseases and receiving immunosuppressive drugs
* kidney transplant recipients
* undergoing hemodialysis or continuous ambulatory peritoneal dialysis
* written informed consent

Exclusion Criteria:

* Allergy to egg proteins
* Former adverse reactions to prior vaccination
* Febrile conditions at the time of study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Immunogenicity defined as seroconversion (1:>=4) and seroprotection rates (1:>=40) | >60 Wochen

SECONDARY OUTCOMES:
Reactogenicity in rheumatologic patients by disease specific scores | Six weeks after vaccination
Immediate side effects at time of application of vaccination | Minutes after vaccination
Side effects after vaccination | First week after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: John M Evison, MD, Principal Investigator — Department of Infectious Diseases, University Hospital Bern, 3010-Bern, Switzerland
Locations (3):
- Switzerland (3):
  - Department of Infectious Diseases, Bern University Hospital, Bern
  - Department of Nephrology/Hypertension, Bern University Hospital, Bern
  - Department of Rheumatic Diseases, Bern University Hospital, Bern

REFERENCES:
- [Background] Vilchez RA, Fung J, Kusne S. The pathogenesis and management of influenza virus infection in organ transplant recipients. Transpl Infect Dis. 2002 Dec;4(4):177-82. doi: 10.1034/j.1399-3062.2002.t01-4-02001.x. PMID 12535259
- [Background] Bridges CB, Fukuda K, Cox NJ, Singleton JA; Advisory Committee on Immunization Practices. Prevention and control of influenza. Recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2001 Apr 20;50(RR-4):1-44. PMID 11334444
- [Background] Kroon FP, van Dissel JT, de Jong JC, van Furth R. Antibody response to influenza, tetanus and pneumococcal vaccines in HIV-seropositive individuals in relation to the number of CD4+ lymphocytes. AIDS. 1994 Apr;8(4):469-76. doi: 10.1097/00002030-199404000-00008. PMID 7912086
- [Background] Dorrell L, Hassan I, Marshall S, Chakraverty P, Ong E. Clinical and serological responses to an inactivated influenza vaccine in adults with HIV infection, diabetes, obstructive airways disease, elderly adults and healthy volunteers. Int J STD AIDS. 1997 Dec;8(12):776-9. doi: 10.1258/0956462971919264. PMID 9433953
- [Background] Chalmers A, Scheifele D, Patterson C, Williams D, Weber J, Shuckett R, Teufel A. Immunization of patients with rheumatoid arthritis against influenza: a study of vaccine safety and immunogenicity. J Rheumatol. 1994 Jul;21(7):1203-6. PMID 7966058
- [Background] Abu-Shakra M, Press J, Varsano N, Levy V, Mendelson E, Sukenik S, Buskila D. Specific antibody response after influenza immunization in systemic lupus erythematosus. J Rheumatol. 2002 Dec;29(12):2555-7. PMID 12465151
- [Background] Cavdar C, Sayan M, Sifil A, Artuk C, Yilmaz N, Bahar H, Camsari T. The comparison of antibody response to influenza vaccination in continuous ambulatory peritoneal dialysis, hemodialysis and renal transplantation patients. Scand J Urol Nephrol. 2003;37(1):71-6. doi: 10.1080/00365590310008749. PMID 12745749
- [Background] Conne P, Gauthey L, Vernet P, Althaus B, Que JU, Finkel B, Gluck R, Cryz SJ Jr. Immunogenicity of trivalent subunit versus virosome-formulated influenza vaccines in geriatric patients. Vaccine. 1997 Oct;15(15):1675-9. doi: 10.1016/s0264-410x(97)00087-x. PMID 9364699
- [Background] Baldo V, Menegon T, Bonello C, Floreani A, Trivello R; Collaborative Group. Comparison of three different influenza vaccines in institutionalised elderly. Vaccine. 2001 May 14;19(25-26):3472-5. doi: 10.1016/s0264-410x(01)00060-3. PMID 11348713
- [Background] Zanetti AR, Amendola A, Besana S, Boschini A, Tanzi E. Safety and immunogenicity of influenza vaccination in individuals infected with HIV. Vaccine. 2002 Dec 20;20 Suppl 5:B29-32. doi: 10.1016/s0264-410x(02)00511-x. PMID 12477415
- [Derived] Evison J, Farese S, Seitz M, Uehlinger DE, Furrer H, Muhlemann K. Randomized, double-blind comparative trial of subunit and virosomal influenza vaccines for immunocompromised patients. Clin Infect Dis. 2009 May 15;48(10):1402-12. doi: 10.1086/598193. PMID 19361304